CLINICAL TRIAL: NCT04505306
Title: Comparison of Short-pulse Subthreshold (532 nm) and Infrared Micropulse (810 nm) Macular Laser for Diabetic Macular Edema
Brief Title: Short-pulse Subthreshold vs Infrared Micropulse for Diabetic Macular Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moorfields Eye Hospital Centre Abu Dhabi (Other)
Collaborators: King Khaled Eye Specialist Hospital (Other Government); University of Nebraska (Other)
Responsible Party: Principal Investigator, Igor Kozak, Consultant Vitreoretinal Surgeon/Clinical Lead, Moorfields Eye Hospital Centre Abu Dhabi
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Moorfields Eye Abu Dhabi
Record Dates: First submitted 2020-08-02; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Diabetic Macular Edema
Keywords: micropulse laser

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subthreshold Laser 30% (Active Comparator): Patients in the SPCW group were treated with grid pattern laser with 20ms pulse PASCAL laser 532nm (TopCon Medical Laser Systems, Tokyo, Japan) with 30% EndPoint algorithm.
  Interventions: Procedure: Macular Laser
- Subtreshold Laser 50% (Active Comparator): Patients in the SPCW group were treated with grid pattern laser with 20ms pulse PASCAL laser 532nm (TopCon Medical Laser Systems, Tokyo, Japan) with 50% EndPoint algorithm.
  Interventions: Procedure: Macular Laser
- Micropulse Laser (Active Comparator): Patients in the STMP group were treated with the 810-nm diode micropulse scanning laser TxCell™ (IRIDEX Corporation, Mountain View, CA, USA) at 15% duty cycle.
  Interventions: Procedure: Macular Laser

INTERVENTIONS:
Procedure: Macular Laser — All treatments were performed using SPCW EndPoint 30% and 50% protocols and STMP laser. Patients in the STMP group were treated with the 810-nm diode micropulse scanning laser TxCell™ (IRIDEX Corporation, Mountain View, CA, USA) at 15% duty cycle. Laser was applied in the confluent mode (low intensity/high density) to cover the entire area of the macular edema and leakage as imaged by OCT and/or fundus fluorescein angiography. Patients in the SPCW group were treated with grid pattern laser with 20ms pulse PASCAL laser 532nm (TopCon Medical Laser Systems, Tokyo, Japan) with EndPoint algorithm, which was either 30% or 50% of testing burn with one burn width apart. In both groups, subthreshold power was determined by titrating burn to light (barely visible) burn and switching to either micropulse mode with 15% duty cycle or 30% and 50% EndPoint value.

SUMMARY:
When applied according to manufacturer recommendations, short-pulse system may yield more temporary reduction in edema while infrared micropulse system may yield slightly better functional outcomes.

DETAILED DESCRIPTION:
Purpose: To assess both anatomic and functional outcomes between short-pulse continuous wavelength and infrared micropulse lasers in the treatment of DME.

Materials and Methods: A prospective interventional study from tertiary care eye hospital - King Khaled Eye Specialist Hospital (Riyadh, Saudi Arabia). Patients with center-involving diabetic macular edema were treated with subthreshold laser therapy. Patients in the micropulse group were treated with the 810-nm diode micropulse scanning laser TxCell™ (IRIDEX Corporation, Mountain View, CA, USA). Laser was applied according to manufacturer recommendations for MicroPulseTM in a confluent mode (low intensity/high density) to the entire area of the macular edema. Patients in the short-pulse group were treated with grid pattern laser with 20ms pulse PASCAL laser 532nm (TopCon Medical Laser Systems, Tokyo, Japan) with EndPoint algorithm, which was either 30% or 50% of testing burn. Main outcome measures included best-corrected visual acuity (BCVA) and foveal thickness at baseline and the last follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* center-involving clinically significant macular edema due to diabetic retinopathy (>300 microns)
* clear ocular media
* ETDRS visual acuity >29 letters (Snellen equivalent of 20/150) or better
* treatment naïve eyes or previously treated with antiangiogenic intravitreal agent(s) more than 6 months ago to allow for long wash-out period

Exclusion Criteria:

* non-center involving diabetic macular edema
* previous retinal laser or surgery
* intravitreal steroid use
* any condition that may be associated with a risk of macular edema such as age-related macular degeneration, retinal vein occlusion, vitreomacular traction, epiretinal membrane and others.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Central foveal thickness | 6 months
  All patients had central retinal thickness measurement using spectral-domain optical coherence tomography (SD-OCT)(Spectralis, Heidelberg Engineering, Heidelberg, Germany). The SD-OCT B-scan was based on the Spectralis macular raster consisting of 19 horizontals 6 millimeter line scans and a real-time eye tracking system.
Best corrected visual acuity | 6 months
  ETDRS visual acuity charts

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfields Eye Hospital Centre, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No